CLINICAL TRIAL: NCT03138655
Title: A Phase 2, Randomized, Double-Blind, Dose-Ranging Study to Determine the Pharmacokinetics, Safety and Tolerability of Vedolizumab IV in Pediatric Subjects With Ulcerative Colitis or Crohn's Disease
Brief Title: Vedolizumab IV in Pediatric Participants With Ulcerative Colitis (UC) or Crohn's Disease (CD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLN0002-2003; 2017-002231-41 (EudraCT Number); U1111-1174-2041 (Other: WHO); MLN0002-2003CTIL (Registry Identifier: Israel); 17/NE/0257 (Registry Identifier: NRES); MOH_2017-09-18_000675 (Other: CRS)
Record Dates: First submitted 2017-04-19; First posted 2017-05-03 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- UC: <30 kg Participants, Vedolizumab 100 mg (Experimental): Participants with UC having baseline weight of <30 kg were randomized to this low dose group and received vedolizumab 100 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- UC: <30 kg Participants, Vedolizumab 200 mg (Experimental): Participants with UC having baseline weight of <30 kg were randomized to this high dose group and received vedolizumab 200 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- CD: <30 kg Participants, Vedolizumab 100 mg (Experimental): Participants with CD having baseline weight of <30 kg were randomized to this low dose group and received vedolizumab 100 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- CD: <30 kg Participants, Vedolizumab 200 mg (Experimental): Participants with CD having baseline weight of <30 kg were randomized to this high dose group and received vedolizumab 200 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- UC: >=30 kg Participants, Vedolizumab 150 mg (Experimental): Participants with UC having baseline weight of >=30 kg were randomized to this low dose group and received vedolizumab 150 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- UC: >=30 kg Participants, Vedolizumab 300 mg (Experimental): Participants with UC having baseline weight of >=30 kg were randomized to this high dose group and received vedolizumab 300 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- CD: >=30 kg Participants, Vedolizumab 150 mg (Experimental): Participants with CD having baseline weight of >=30 kg were randomized to this low dose group and received vedolizumab 150 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab
- CD: >=30 kg Participants, Vedolizumab 300 mg (Experimental): Participants with CD having baseline weight of >=30 kg were randomized to this low dose group and received vedolizumab 300 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion.
  Other Names: MLN0002; ENTYVIO; KYNTELES

SUMMARY:
The purpose of this study is to evaluate vedolizumab pharmacokinetics (PK), safety and tolerability in pediatric participants with moderately to severely active UC or CD.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat pediatric participants who have moderately to severely active UC or CD. This study will look at the PK, efficacy, immunogenicity, safety, and tolerability in participants who take vedolizumab.

The study will enroll approximately 80 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two dose regimens (high or low) per weight group >=30 kg and 10 kg to <30 kg in ratio 1:1-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Vedolizumab high dose group - Vedolizumab 300 mg or 200 mg
* Vedolizumab low dose group - Vedolizumab 150 mg or 100 mg

All participants will be administered vedolizumab via IV infusion. Participants assigned to the low dose group who do not achieve clinical response (based on pediatric UC/CDAI) at Week 14 will receive the high dose (that is, 300 mg for participants >=30 kg baseline weight and 200 mg for participants 10 kg to <30 kg baseline weight) of vedolizumab IV at Week 14. Participants assigned to the high dose group who had not achieved clinical response continued on the same blinded high dose at Week 14.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 36 weeks. After completing the Week 22 Visit procedures, eligible participants may enter a blinded extension study. Participants will make multiple visits to the clinic, and those who do not enter extension study will have a final visit 18 weeks after last dose of study drug for a follow-up assessment. Participants who do not enter the extension study will also participate in a long-term safety follow-up, by telephone, 6 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participants weighs >=10 kg at the time of randomization.
2. Has a medical history of moderately to severely active UC during Screening defined as complete Mayo score of 6 to 12, and a total Mayo subscores of stool frequency and rectal bleeding >=4 and Mayo endoscopy subscore >=2, or has moderately to severely active CD defined as simple endoscopic score for Crohn's disease (SES-CD) >=7, and the CDAI components of average daily abdominal pain score of greater than (>) 1 for the 7 days prior, and total number of liquid/very soft stools >10 within 7 days prior to first dose of study drug.
3. Has evidence of UC extending proximal to the rectum (that is, not limited to proctitis) or evidence of CD involving the ileum and/or colon, at a minimum.
4. Has extensive colitis or pancolitis of >8 years duration or left-sided colitis of >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months prior to their first dose of study drug.
5. Has a family history of colorectal cancer (that is, first-degree relative), personal history of increased colorectal cancer risk, or other known risk factor must be up-to-date on colorectal cancer surveillance.
6. The participant's vaccinations are up to date.
7. Has demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents as defined below:

   Corticosteroids:

   • Signs and/or symptoms of persistently active disease despite a history of at least one 4-week induction regimen that included a dose equivalent to or more than prednisone 1 milligram per kilogram (mg/kg) daily orally for 2 weeks or IV for 1 week.

   OR

   • Two failed attempts to taper corticosteroids to below a dose equivalent to prednisone 10 mg daily orally on 2 separate occasions.

   OR

   • History of significant intolerance to corticosteroids (including, but not limited to, Cushing's syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, and infection).

   Immunomodulators:

   • Signs and symptoms of persistently active disease despite a history of at least one 8-week regimen of oral azathioprine (AZA) (>=1.5 milligram per kilogram per day [mg/kg/day]) or 6-mercaptopurine (6-MP) mg/kg (>=1.0 mg/kg/day) or methotrexate (MTX) (>=10 milligram per square meter [mg/m^2] once a week).

   OR

   • History of intolerance of at least 1 immunomodulator (including, but not limited to, nausea/vomiting, abdominal pain, pancreatitis, liver function test (LFT) abnormalities, lymphopenia, thiopurine methyltransferase genetic mutation, infection).

   Tumor necrosis factor-alpha (TNF-α) antagonists:

   • Signs and symptoms of persistently active disease despite a history of at least 1 induction regimen of infliximab 5 mg/kg IV at Week 0 and Weeks 2 and 6 or adalimumab 2-week regimen of 160 mg on Day 1 and 80 mg on Day 15 if >=40 kg or 80 mg on Day 1 and 40 mg on Day 15 if <40 kg. For any other TNF-α antagonist, the participant must demonstrate signs and symptoms of persistently active disease despite a history of at least 1 induction regimen, as determined by the investigator.

   OR

   • Recurrence of symptoms during maintenance dosing following prior clinical benefit, that is, fitting clinically with secondary loss of response (discontinuation despite clinical benefit does not qualify).

   OR

   • History of intolerance of infliximab or adalimumab (including, but not limited to, infusion-related reaction, demyelination, congestive heart failure, infection).
8. The participant may be receiving a therapeutic dose of the following drugs:

   1. Oral 5-aminosalicylic acid (5-ASA) compounds, providing the dose has been stable for the 2 weeks prior to first dose of study drug.
   2. Oral corticosteroid therapy (prednisolone at a stable dose <=50 mg/day, or equivalent steroid), provided that the dose has been stable for the 4 weeks prior to first dose of study drug if corticosteroids have been initiated, or for the 2 weeks prior to first dose of study drug if corticosteroids are being tapered.
   3. Probiotics (example, Saccharomyces boulardii), provided the dose has been stable for the 2 weeks prior to first dose of study drug.
   4. Antidiarrheals (example, loperamide, diphenoxylate with atropine) for control of chronic diarrhea.
   5. Antibiotics used for the treatment of CD (example, ciprofloxacin, metronidazole), providing the dose has been stable for the 2 weeks prior to first dose of study drug.
   6. Azathioprine or 6-MP, provided the dose has been stable for the 8 weeks prior to first dose of study drug.
   7. Methotrexate (MTX), provided the dose has been stable for the 8 weeks prior to first dose of study drug.

Exclusion Criteria:

1. Has had previous exposure to approved or investigational anti-integrins (example, natalizumab, efalizumab, etrolizumab, or AMG 181) or MAdCAM-1 antagonists, or rituximab.
2. Has had prior exposure to vedolizumab.
3. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist prior to the administration of the first dose of study drug.
4. Requires surgical intervention for UC or CD, or is anticipated to require surgical intervention for UC or CD during this study.
5. Use of topical (rectal) treatment with 5-ASA or corticosteroid enemas/suppositories within 2 weeks of the administration of the first dose of study drug.
6. Has any unstable or uncontrolled cardiovascular, heart failure moderate to severe (New York Class Association III or IV), pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, coagulation, immunological, endocrine/metabolic, neurological, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
7. Active or latent tuberculosis (TB), as evidenced by a diagnostic TB test performed within 30 days of Screening or during the Screening Period that is positive, defined as:

   * Positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR
   * A TB skin test reaction >=5 millimeter (mm). Participants with documented previously treated TB with a negative QuantiFERON test can be included in the study.
8. Clinically significant current or recent history (within 1 year prior to enrollment) of alcohol dependence or illicit drug use.
9. Has a current diagnosis of indeterminate colitis (Inflammatory bowel disease unclassified [IBDU]). For participants less than 6 years of age, any findings that suggest monogenic very early onset inflammatory bowel disease should be excluded.
10. Has evidence of abdominal abscess or toxic megacolon at the initial Screening Visit.
11. Has ileostomy, colostomy, ileo-anal pouch, or known fixed symptomatic stenosis of the intestine.
12. Has extensive colonic resection, example, subtotal or total colectomy.
13. Has a history or evidence of adenomatous colonic polyps that have not been removed.
14. Has a history or evidence of colonic mucosal dysplasia.
15. Has chronic hepatitis B virus (HBV) infection* or chronic hepatitis C virus (HCV) infection. * HBV immune participants (that is, being hepatitis B surface antigen [HBsAg] negative and hepatitis B antibody positive) may be included, however.
16. Has any identified congenital or acquired immunodeficiency (example, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
17. Has evidence of or treatment for Clostridium difficile (C difficile) infection within 60 days or other intestinal pathogen within 30 days prior to first dose of study drug.
18. Has any history of malignancy, except for the following: (a) adequately treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to enrollment; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to first dose of study drug. Participants with remote history of malignancy (example, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received, and inclusion must be discussed with the sponsor on a case-by-case basis prior to enrollment.
19. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
20. Has history of lupus.
21. Has had a surgical procedure requiring general anesthesia within 30 days prior to screening or is planning to undergo major surgery during the study period.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Science, Study Director — Takeda
Locations (88):
- United States (27):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Wilmington, Delaware
  - Nemours Childrens Specialty Care - Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University School of Medicine - Indianapolis, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Northwell Health, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Childrens Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Specialty Group - Medical Center Location, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Belgium (4):
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre University Hospital, London, Ontario
  - Toronto Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre Glen Site, Montreal, Quebec
- France (4):
  - Hopital Jeanne de Flandre, Lille, Hauts-de-France
  - Hopital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital Necker-Enfants Malades, Paris, Île-de-France Region
  - Hopital Robert Debre, Paris, Île-de-France Region
- Germany (5):
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Ludwig-Maximillians-Universitat Munchen, München, Bavaria
  - Universitatsmedizin Rostock - Kinder und Jugendklinik, Rostock, Mecklenburg-Vorpommern
  - Universitatsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
- Hungary (5):
  - BAZ Megyei Korhaz es Egyetemi Oktatokorhaz, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet, Sopron, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem, Budapest
- Israel (8):
  - Soroka University Medical Center, Beersheba, Beersheba
  - Schneider Children's Medical Center of Israel, Petach Tikvah, Petah Tiqwa
  - Assaf Harofeh Medical Center, Ẕerifin, Rehoboth
  - The Edmond and Lily Safra Children's Hospital - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (4):
  - Radboud Universitair Medisch Centrum, Nijmegen, GA
  - Emma Kinderziekenhuis AMC, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel
  - Erasmus University Medical Center, Rotterdam, South Holland
- Poland (9):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Warszawski Uniwersytet Medyczny, Warsaw, Masovian Voivodeship
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów, Podkarpackie Voivodeship
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Copernicus Podmiot Leczniczy, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Specjalistyczny Zaklad Opieki Zdrowotnej ZDROJE, Szczecin, West Pomeranian Voivodeship
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi Osrodek Pediatryczny im Marii Konopnic, Lodz, Łódź Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Ukraine (2):
  - National Scientific Center of Radiological Medicine of NAMS of Ukraine, Kyiv, KIEV CITY
  - Kharkiv Regional Clinical Children's Hospital, Kharkiv
- United Kingdom (10):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, England
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Barts and The London NHS Trust, London, England
  - King's College Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - Sheffield Children's NHS Foundation Trust, Sheffield, England
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 72 investigative sites in United States, Belgium, Canada, France, Germany, Hungary, Israel, Netherlands, Poland, Ukraine, United Kingdom and European Union from 8 November 2017 to 26 March 2020.
Pre-assignment Details: Pediatric participants who weighed >10 kg with a diagnosis of moderately to severely active ulcerative colitis (UC) or Crohn's disease (CD) were enrolled in 1:1 ratio to receive vedolizumab low or high dose groups per weight (<30 kg and >=30 kg).
Period: Overall Study
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg
Started | 10 | 9 | 11 | 10 | 13 | 12 | 12 | 12
Completed | 7 | 7 | 9 | 7 | 11 | 7 | 9 | 10
Not Completed | 3 | 2 | 2 | 3 | 2 | 5 | 3 | 2
Not completed — Adverse Event | 2 | 1 | 2 | 1 | 1 | 4 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason not Specified | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who are randomized into the study regardless whether they received any dose of study drug or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg | Total
Number analyzed (Participants) | 10 | 9 | 11 | 10 | 13 | 12 | 12 | 12 | 89
Age, Continuous [Mean (Full Range); unit: years] | 7.0 [3 to 12] | 8.0 [2 to 12] | 7.4 [2 to 12] | 8.1 [3 to 12] | 12.4 [8 to 17] | 13.9 [9 to 17] | 13.4 [10 to 17] | 14.3 [11 to 17] | 10.56 [2 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 5 | 5 | 6 | 8 | 3 | 39
  Male | 6 | 5 | 7 | 5 | 8 | 6 | 4 | 9 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 9
  Not Hispanic or Latino | 10 | 7 | 7 | 8 | 12 | 11 | 11 | 12 | 78
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 8
  White | 7 | 7 | 7 | 9 | 11 | 10 | 9 | 11 | 71
  More than one race | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 5
  France | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Hungary | 1 | 0 | 1 | 1 | 3 | 4 | 4 | 3 | 17
  Poland | 2 | 1 | 4 | 2 | 1 | 0 | 2 | 3 | 15
  United Kingdom | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 6
  Ukraine | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Israel | 3 | 2 | 0 | 2 | 3 | 2 | 0 | 1 | 13
  Canada | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  United States | 2 | 5 | 4 | 4 | 5 | 5 | 2 | 2 | 29
Height [Mean (Full Range); unit: cm] | 119.59 [82.7 to 146.0] | 122.39 [84.9 to 143.0] | 120.58 [83.5 to 146.0] | 124.67 [96.5 to 137.6] | 153.11 [128.0 to 176.1] | 160.03 [138.3 to 185.4] | 157.85 [134.3 to 182.5] | 157.98 [141.9 to 181.5] | 139.53 [82.7 to 185.4]
Weight [Mean (Full Range); unit: kg] | 22.38 [12.8 to 29.6] | 23.23 [10.2 to 29.8] | 22.06 [12.0 to 29.9] | 23.37 [14.3 to 30.0] | 46.22 [30.3 to 75.9] | 53.98 [32.0 to 78.9] | 51.53 [31.4 to 79.0] | 45.89 [33.9 to 68.0] | 36.08 [10.2 to 79.0]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — BMI = weight (kg) / height^2 (m^2)
  kg/m^2 | 15.63 [13.4 to 18.7] | 15.29 [12.4 to 20.0] | 15.04 [13.5 to 17.2] | 14.93 [12.4 to 16.9] | 19.51 [16.4 to 26.5] | 20.76 [16.7 to 27.1] | 20.50 [14.4 to 24.5] | 18.26 [15.8 to 25.9] | 17.49 [12.4 to 27.1]

OUTCOME MEASURES:

1. Primary Outcome: AUCWeek 14: Area Under the Serum Concentration-time Curve at Week 14
Time Frame: From Day 43 (Week 6) post-dose up to pre-dose Day 99 (Week 14)
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least 1 dose of study drug and had at least 1 measurable concentration of vedolizumab. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 11 | 10 | 9 | 10
h*ng/mL | 1933.5076 (1184.36284) | 3231.1001 (1152.06628) | 2344.4204 (1216.58345) | 3091.7957 (1732.34795) | 2449.9433 (772.66677) | 4182.4869 (1751.87940) | 1865.0004 (509.68268) | 3176.6971 (928.32630)

2. Primary Outcome: Cav,Week 14: Average Serum Concentration During a Dosing Interval at Week 14
Time Frame: From Day 43 (week 6) post-dose up to pre-dose Day 99 (Week 14)
Population: PK Analysis Set included all participants who received at least 1 dose of study drug and had at least 1 measurable concentration of vedolizumab. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg
Number analyzed (Participants) | 9 | 8 | 7 | 8 | 11 | 10 | 9 | 10
ng/mL | 39.3143 (21.34097) | 61.2934 (18.14446) | 46.8716 (23.07334) | 63.6275 (28.29116) | 44.6465 (11.48500) | 77.2452 (28.49511) | 37.4752 (18.26528) | 63.1734 (15.08119)

3. Primary Outcome: Ctrough,Week 14: Observed Serum Concentration at the End of a Dosing Interval at Week 14
Time Frame: At the end of a dosing interval at Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 11 | 10 | 10 | 10
ng/mL | 9.3100 (9.48045) | 10.7226 (10.35423) | 8.7395 (7.77386) | 10.3685 (11.30124) | 16.3645 (16.93869) | 21.4860 (18.01872) | 3.9006 (3.62991) | 7.8310 (9.44044)

4. Secondary Outcome: Percentage of UC Participants Who Achieve Clinical Response Based on Complete Mayo Score
Description: Clinical response was defined as a reduction in complete Mayo score of >= 3 points and >=30 % from Baseline with an accompanying decrease in rectal bleeding sub-score of >=1 point(s) or absolute rectal bleeding sub-score of <= 1 point. Mayo score was used in to assess UC disease activity. It consisted of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale was scored on a scale of 0 to 3, where 0= normal condition and 3 = severe disease condition. The total Mayo score ranged from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Baseline (Day 1) and Week 14
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UC: <30 kg Participants, Vedolizumab 100 mg | UC: <30 kg Participants, Vedolizumab 200 mg | UC: >=30 kg Participants, Vedolizumab 150 mg | UC: >=30 kg Participants, Vedolizumab 300 mg
Number analyzed (Participants) | 10 | 9 | 13 | 12
percentage of participants | 40.0 [12.2 to 73.8] | 66.7 [29.9 to 92.5] | 69.2 [38.6 to 90.9] | 41.7 [15.2 to 72.3]

5. Secondary Outcome: Percentage of CD Participants Who Achieve Clinical Response Based on Crohn's Disease Activity Index (CDAI)
Description: Clinical response was defined as >=70 points decrease from Baseline in CDAI score at Week 14. The CDAI evaluated severity of signs and symptoms of CD. Information was collected on number of liquid stools, intensity of abdominal pain, general well-being, presence of comorbid conditions, use of medications for diarrhea, physical examination, and laboratory, yielding 8 items that were combined with data from a 7-day diary to obtain total CDAI score. Index values of 150 and below were associated with quiescent disease; values above that indicated active disease, values >=220 indicated moderate to severe disease, and values above 450 were seen with extremely severe disease.
Time Frame: Baseline (Day 1) and Week 14
Population: FAS included all randomized participants who received at least 1 dose of study drug. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD: <30 kg Participants, Vedolizumab 100 mg | CD: <30 kg Participants, Vedolizumab 200 mg | CD: >=30 kg Participants, Vedolizumab 150 mg | CD: >=30 kg Participants, Vedolizumab 300 mg
Number analyzed (Participants) | 11 | 10 | 11 | 12
percentage of participants | 63.6 [30.8 to 89.1] | 40.0 [12.2 to 73.8] | 45.5 [16.7 to 76.6] | 33.3 [9.9 to 65.1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 32
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included all participants who received at least 1 dose of study drug. MedDRA v22.0 was used for >30 kg group and v23.0 for <30 kg group).
Groups:
- <30 kg Participants, Vedolizumab 100 mg: Participants with UC or CD having baseline weight of <30 kg, were randomized to this low dose group and received vedolizumab 100 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
- <30 kg Participants, Vedolizumab 200 mg: Participants with UC or CD having baseline weight of <30 kg, were randomized to this high dose group and received vedolizumab 200 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
- <30 kg Participants, Vedolizumab 100 mg to 200 mg: Participants from '<30 kg Participants, Vedolizumab 100 mg' low dose group who did not achieve Clinical Response at Week 14 were escalated to receive vedolizumab 200 mg IV infusion at Week 14.
- >=30 kg Participants, Vedolizumab 150 mg: Participants with UC or CD having baseline weight of >=30 kg, were randomized to this low dose group and received vedolizumab 150 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
- >=30 kg Participants, Vedolizumab 300 mg: Participants with UC or CD having baseline weight of >=30 kg, were randomized to this low dose group and received vedolizumab 300 mg IV infusion on Day 1 and at Weeks 2, 6 and 14.
- >=30 kg Participants, Vedolizumab 150 mg to 300 mg: Participants from '>=30 kg Participants, Vedolizumab 150 mg' low dose group who did not achieve Clinical Response at Week 14 were escalated to receive vedolizumab 300 mg IV infusion at Week 14.
Arm/Group | <30 kg Participants, Vedolizumab 100 mg | <30 kg Participants, Vedolizumab 200 mg | <30 kg Participants, Vedolizumab 100 mg to 200 mg | >=30 kg Participants, Vedolizumab 150 mg | >=30 kg Participants, Vedolizumab 300 mg | >=30 kg Participants, Vedolizumab 150 mg to 300 mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19 | 0/4 | 0/18 | 0/24 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/17 | 6/19 | 2/4 | 2/18 | 8/24 | 1/6
Other Adverse Events (participants affected / at risk) | 16/17 | 13/19 | 3/4 | 15/18 | 20/24 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | <30 kg Participants, Vedolizumab 100 mg (N=17) | <30 kg Participants, Vedolizumab 200 mg (N=19) | <30 kg Participants, Vedolizumab 100 mg to 200 mg (N=4) | >=30 kg Participants, Vedolizumab 150 mg (N=18) | >=30 kg Participants, Vedolizumab 300 mg (N=24) | >=30 kg Participants, Vedolizumab 150 mg to 300 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | <30 kg Participants, Vedolizumab 100 mg (N=17) | <30 kg Participants, Vedolizumab 200 mg (N=19) | <30 kg Participants, Vedolizumab 100 mg to 200 mg (N=4) | >=30 kg Participants, Vedolizumab 150 mg (N=18) | >=30 kg Participants, Vedolizumab 300 mg (N=24) | >=30 kg Participants, Vedolizumab 150 mg to 300 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 3 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1
Viral infection (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 1
Clostridium test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Torus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 3 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fear of injection (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03138655/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT03138655/SAP_001.pdf